CLINICAL TRIAL: NCT06733038
Title: Phase III Randomized Study of FOLFOXIRI Plus Bevacizumab and Atezolizumab Versus FOLFOXIRI Plus Bevacizumab as First-Line Treatment of Unresectable pMMR and Immunoscore IC-High Metastatic Colorectal Cancer Patients
Brief Title: FOLFOXIRI Plus Bevacizumab With or Without Atezolizumab as 1st Line Treatment of pMMR and IS IC-High Metastatic Colorectal Cancer Patients.
Acronym: AtezoTRIBE2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AtezoTRIBE2
Record Dates: First submitted 2024-12-02; First posted 2024-12-13 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
Keywords: atezolizumab; FOLFIXIRI/bevacizumab; metastatic colorectal cancer; pMMR/MSS; IMMUSCORE IC-High; first line
MeSH Terms: conditions — Colorectal Neoplasms | interventions — atezolizumab; Bevacizumab; Irinotecan; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - FOLFOXIRI plus bevacizumab (Active Comparator): Every 2 weeks for a maximum of 8 cycles:
  * Bevacizumab 5 mg/kg iv 90 minutes at cycle 1 (if well tolerated, it is administered over 60 minutes at cycle 2, and over 30 minutes at cycle 3) day 1, followed by
  * Irinotecan 165 mg/sqm iv over 60 minutes day 1, followed by
  * Oxaliplatin 85 mg/sqm iv over 2 hours day 1, in two-way with
  * L-Leucovorin 200 mg/sqm iv over 2 hours day 1, followed by
  * 5-fluorouracil 3200 mg/sqm 48 h-continuous infusion, starting on day 1.
  If no progression occurs during FOLFOXIRI plus bev, patients will receive maintenance 5-FU/LV plus bev at the same dose used at the last cycle of the induction treatment. 5-FU/LV plus bev will be repeated biweekly until disease progression, unacceptable toxicity or patient's refusal.
  Interventions: Drug: Bevacizumab; Drug: Irinotecan (CPT-11); Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil (5-FU)
- Arm B - FOLFOXIRI plus bevacizumab plus atezolizumab (Experimental): Every 2 weeks for a maximum of 8 cycles:
  * Atezolizumab 840 mg iv over 30 minutes (60 minutes at first infusion) day 1 followed by
  * Bevacizumab 5 mg/kg iv over 90 minutes at cycle 1 (if well tolerated, it is administered over 60 minutes at cycle 2, and over 30 minutes at cycle 3) day 1 followed by
  * Irinotecan 165 mg/sqm iv over 60 minutes day 1, followed by
  * Oxaliplatin 85 mg/sqm iv over 2 hours day 1, in two-way with
  * L-Leucovorin 200 mg/sqm iv over 2 hours day 1, followed by
  * 5-fluorouracil 3200 mg/sqm 48 h-continuous infusion, starting on day 1.
  If no progression occurs during FOLFOXIRI plus bev plus atezolizumab, patients will receive maintenance 5-FU/LV plus bev plus atezolizumab at the same dose used at the last cycle of the induction treatment. 5-FU/LV plus bev plus atezolizumab will be repeated biweekly until disease progression, unacceptable toxicity or patient's refusal.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Irinotecan (CPT-11); Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil (5-FU)

INTERVENTIONS:
Drug: Atezolizumab — 840 mg iv over 30 minutes (60 minutes at first infusion) day 1
  Arms: Arm B - FOLFOXIRI plus bevacizumab plus atezolizumab
Drug: Bevacizumab — 5 mg/kg iv over 90 minutes at cycle 1 (if well tolerated, it is administered over 60 minutes at cycle 2, and over 30 minutes at cycle 3) day 1
Drug: Irinotecan (CPT-11) — 165 mg/sqm iv over 60 minutes day 1
Drug: Oxaliplatin — 85 mg/sqm iv over 2 hours day 1
Drug: Leucovorin — 200 mg/sqm iv over 2 hours day 1
Drug: Fluorouracil (5-FU) — 3200 mg/sqm 48 h-continuous infusion, starting on day 1

SUMMARY:
The aim of this study is to evaluate the efficacy of the addition of Atezolizumab to FOLFOXIRI plus bevacizumab as first line treatment of patients with pMMR and Immunoscore IC-high metastatic colorectal cancer in terms of Progression Free Survival (PFS).

DETAILED DESCRIPTION:
This is a prospective, open-label, multicenter phase III randomized trial in which patients with initially unresectable, previously untreated pMMR and Immunoscore IC-high mCRC will be randomized in a 1:1 ratio to receive induction treatment with FOLFOXIRI plus bevacizumab up to 8 cycles followed by maintenance with 5-FU/LV plus bevacizumab until disease progression, unacceptable toxicity or patient's refusal (arm A) or FOLFOXIRI plus bevacizumab plus atezolizumab up to 8 cycles followed by maintenance with 5-FU/LV plus bevacizumab plus atezolizumab until disease progression, unacceptable toxicity or patient's refusal (arm B).

Stratification factors will be ECOG Performance Status (0 versus 1, 2), primary tumour location (right versus left/rectum) and liver metastases (yes versus no).

The second- and subsequent lines of treatment will be at investigators' choice.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of colorectal cancer;
* Initially unresectable metastatic colorectal cancer not previously treated with chemotherapy for metastatic disease;
* Proficient mismatch repair (pMMR) status in tumour tissue (primary or metastatic), as determined by a local laboratory assay in a CLIA- or similarly certified;
* Immunoscore IC-high status in tumour tissue (primary or metastatic), as determined by a sponsor-defined central laboratory (HEGP, AP-HP, INSERM, France).
* At least one measurable lesion according to RECIST criteria (version 1.1);
* Availability of adequate tumour specimen (primary or metastatic);
* Male or female of 18-75 years of age;
* ECOG PS ≤ 2 if aged < 71 years, ECOG PS = 0 if aged 71-75 years;
* Life expectancy of at least 12 weeks;
* Previous adjuvant chemotherapy allowed only if with fluoropyrimidine monotherapy and more than 6 months elapsed between the end of adjuvant and first relapse;
* Neutrophils >1.5 x 109/L, Platelets >100 x 109/L, Hb >9 g/dl;
* Total bilirubin ≤1.5 times the upper-normal limits (UNL) of the normal values and AST (SGOT) and/or ALT (SGPT) <2.5 x UNL (or <5 x UNL in case of liver metastases) alkaline phosphatase <2.5 x UNL (or <5 x UNL in case of liver metastases);
* Creatinine clearance ≥50 mL/min or serum creatinine ≤1.5 x UNL;
* INR or aPTT ≤1.5 x ULN. This applies only to patients who are not receiving therapeutic anticoagulation;
* Urine dipstick of proteinuria <2+. Patients discovered to have 2+ proteinuria on dipstick urinalysis at baseline, should undergo a 24-hour urine collection and must demonstrate ≤1 g of protein/24 h;
* Women of childbearing potential must have a negative blood pregnancy test at the baseline visit. For this trial, women of childbearing potential are defined as all women following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient;
* Male subjects with female partners of childbearing potential and female subjects of childbearing potential must, therefore, be willing to use adequate contraception as approved by the investigator (barrier contraceptive measure or oral contraception) and outlined in "Section 6.5 - Contraception", starting with the first dose of study therapy through 6 months after the last dose of bevacizumab and fluorouracil and within 5 months after the last dose of atezolizumab.
* Females of childbearing potential must have a negative blood pregnancy test at the baseline visit (i.e., performed maximum 7 days before the treatment start);
* Will and ability to comply with the protocol;
* Written informed consent to study procedures.

Exclusion Criteria:

* Radiotherapy to any site within 4 weeks before the study;
* Previous adjuvant oxaliplatin-containing chemotherapy;
* Previous treatment with bevacizumab;
* Prior treatment with CD137 agonists, anti-CTLA4, anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents;
* Complete dihydropyrimidine dehydrogenase (DPYD) deficiency (homozygous of the following DPYD polymorphisms: c1679GG, c1905+1AA, c2846TT);
* Untreated brain metastases or spinal cord compression or primary brain tumours;
* History or evidence upon physical examination of CNS disease unless adequately treated;
* History of haemoptysis ≥ 2 grade NCIC-CTG criteria within one month prior to screening;
* Active or untreated CNS metastases:
* Symptomatic peripheral neuropathy > 2 grade NCIC-CTG criteria;
* Serious, non-healing wound, ulcer, or bone fracture;
* Evidence of bleeding diathesis or coagulopathy;
* Uncontrolled hypertension (SBP>150 mmHg and/or DPB>100 mmHg), or prior history of hypertensive crisis, or hypertensive encephalopathy ;
* Clinically significant (i.e., active) cardiovascular disease for example cerebrovascular accidents (within 6 months prior to study enrollment), myocardial infarction (within 6 months prior to study enrollment), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication;
* Significant vascular disease (e.g. aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months of study enrolment;
* Active infection requiring antibiotics at the time of initiation of study treatment;
* Any previous venous thromboembolism ≥ NCI CTCAE Grade 4;
* History of abdominal fistula, GI perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to the first study treatment;
* Current or recent (within 10 days prior to study treatment start) ongoing treatment with full-dose anticoagulants for therapeutic purposes.
* Chronic, daily treatment with high-dose aspirin (>325 mg/day);
* Treatment with any investigational drug within 30 days prior to enrollment or 2 investigational agent half-lives (whichever is longer);
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of localized basal and squamous cell carcinoma or cervical cancer in situ;
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study;
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to initiation of study treatment;
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication;
* Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Sexually active males and females (of childbearing potential) unwilling to practice contraception (barrier contraceptive measure or oral contraception) during the study and until 6 months after the last dose of bevacizumab, fluorouracil and within 5 months after the last dose of atezolizumab;
* History of autoimmune disease;
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan;
* Positive test for human immunodeficiency virus (HIV);
* Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test prior to randomization) or hepatitis C;
* Active tuberculosis;
* Prior allogenic bone marrow transplantation or solid organ transplant;
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumour necrosis factor [TNF] agents) within 2 weeks prior to start of study treatment, or requirement for systemic immunosuppressive medications during the trial. The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed;
* Known hypersensitivity or allergy to Chinese hamster ovary cell products or any component of the atezolizumab formulation;
* Administration of a live, attenuated vaccine within 4 weeks prior to start of study treatment or anticipation that such a live attenuated vaccine will be required during the study;
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin-2) within 4 weeks or five half-lives of the drug, whichever is longer, prior to start of study treatment; • If receiving a RANKL inhibitor (e.g. denosumab), unwilling to adopt alternative treatment such as (but not limited to) bisphosphonates, while receiving atezolizumab.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 24 months
  PFS is defined as the time from randomization to the first documentation of objective disease progression or death due to any cause, whichever occurs first. PFS will be censored on the date of the last evaluable on study tumor assessment documenting absence of progressive disease for patients who are alive, on study and progression free at the time of the analysis. Alive patients having no tumor assessments after baseline will have time to event censored on the date of randomization.

SECONDARY OUTCOMES:
Overall Toxicity Rate | 24 months
  Overall Toxicity Rate is defined as the percentage of patients, relative to the total of enrolled subjects, experiencing any adverse event, according to National Cancer Institute Common Toxicity Criteria (version 5.0), during the induction and the maintenance phases of treatment.
Toxicity Rate | 24 months
  Toxicity Rate is defined as the percentage of patients, relative to the total of enrolled subjects, experiencing a specific adverse event of grade 3/4, according to National Cancer Institute Common Toxicity Criteria (version 5.0), during the induction and the maintenance phases of treatment.
Objective Response Rate | 24 months
  Objective Response Rate (ORR) is defined as the percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria, during the induction and the maintenance phases of treatment. The determination of clinical response will be based on investigator reported measurements. Responses will be evaluated every 8 weeks.
Immuno-related Objective Response Rate | 24 months
  Immuno-related Objective Response Rate (irORR) is defined as the percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to immune-modified RECIST criteria, during the induction and the maintenance phases of treatment. The determination of clinical response will be based on investigator reported measurements. Responses will be evaluated every 8 weeks.
Early Objective Response Rate | up to 2 months from randomization
  Early Objective Response Rate (EOR) is defined as the percentage of patients, relative to the total of the enrolled subjects, achieving a ≥20% decrease in the sum of diameters of RECIST target lesions at week 8 compared to baseline.
Depth of Response | 24 months
  Depth of Response (DpR) is defined as the relative change in the sum of longest diameters of RECIST target lesions at the nadir, in the absence of new lesions or progression of non-target lesions, when compared with baseline.
R0 Resection Rate | 24 months
  R0 Resection Rate is defined as the percentage of patients, relative to the total of enrolled subjects, undergoing secondary R0 resection of metastases. Secondary R0 surgery is defined as microscopically margin free complete surgical removal of all residual disease, performed during treatment or after its completion, allowed by tumoral shrinkage and/or disappearance of one or more lesions.
Duration of Response | 24 months
  Duration of Response (DoR) is defined as the time from first documentation of objective response (complete [CR] or partial [PR] response, per RECIST 1.11) to the first documentation of PD (per RECIST 1.1) or to death to any cause, whichever comes first.
Overall survival | 48 months
  Overall survival (OS) is defined as the time from randomization to the date of death due to any cause. For patients still alive at the time of analysis, the OS time will be censored on the last date the patients were known to be alive.
Quality of Life as assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Questionnaires will be administered at baseline, every 4 weeks during induction treatment, every 8 weeks thereafter, at the time of evidence of disease progression, after 30 days following end of study treatment/disease progression.
  The EORTC QLQ-C30 contains functional scales, symptom scales, single items scale and a global health status/QoL scale. Raw scores are standardized and converted into scale scores ranging from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales. Quality of life will be evaluated for patients who will have completed at least one questionnaire item at baseline and during the study period through descriptive summary statistics.
Quality of Life as assessed by the European Organization for Research and Treatment of Cancer Quality of Life Module for Colorectal cancer 29 (EORTC QLQ-CR29). | Questionnaires will be administered at baseline, every 4 weeks during induction treatment, every 8 weeks thereafter, at the time of evidence of disease progression, after 30 days following end of study treatment/disease progression.
  The EORTC QLQ-CR29 includes 29 items that evaluate symptoms (gastrointestinal, urinary, pain and others) and functional areas (sexual, body image and others) that are associated with CRC and its treatments. There are separate items for patients with and without a stoma and separate items to evaluate the sexual function of men and women. Raw scores are standardized and converted into scale scores ranging from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales. Quality of life will be evaluated for patients who will have completed at least one questionnaire item at baseline and during the study period through descriptive summary statistics.
Time To Deterioration in Quality of Life (TTD) | 24 months
  The time from baseline to the first onset of a 10-point or greater decrease from baseline for functional scales or a 10-point or greater increase for symptom scales or death.

CONTACTS AND LOCATIONS:
Overall Officials: Carlotta Antoniotti, MD, PhD, Principal Investigator — Department of Translational Research and New Technologies in Medicine and Surgery - University of Pisa
Locations (24):
- Italy (24):
  - Fondazione Poliambulanza, Istituto Ospedaliero, Brescia, BS
  - Azienda Ospedaliero Universitaria Policlinico Rodolico - S. Marco, Catania, CT
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori, Meldola, FC
  - Fondazione Casa Sollievo della Sofferenza, San Giovanni Rotondo, FG
  - AOU Careggi, Florence, FI
  - Azienda Ospedaliera Card. G. Panico, Tricase, LE
  - Azienda USL Toscana Nord Ovest, Livorno, LI
  - Ospedale San Luca, Lucca, LU
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, MI
  - Ospedale San Raffaele, Milan, MI
  - Fondazione IRCCS INT - Milano, Milan, MI
  - Azienda Ospedaliero Universitaria di Modena, Modena, MO
  - Istituto Oncologico Veneto Irccs, Padua, PD
  - IRCCS Centro di Riferimento Oncologico, Aviano, PN
  - Nuovo Ospedale di Prato S. Stefano, Prato, PO
  - Azienda USL della Romagna, Ravenna, RA
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, RM
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine, UD
  - ASL di Viterbo, Viterbo, VT
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli, Naples
  - IRCCS Istituto Nazionale Tumori "Fondazione Giovanni Pascale", Napoli
  - Azienda Usl di Piacenza, Piacenza
  - U.O. Oncologia Medica 2 Universitaria - Azienda Ospedaliero-Universitaria Pisana Dipartimento di Ricerca Traslazionale e Nuove Tecnologie - University of Pisa, Pisa
  - Policlinico Universitario Tor Vergata, Rome

IPD SHARING:
Plan to Share IPD: No